CLINICAL TRIAL: NCT06183320
Title: Can Flowable Bulk Fill Composites be Used in Proximal Area of Class II Restorations: A Double-blinded Randomized Clinical Trial
Brief Title: Can Flowable Bulk Fill Composites be Used in Proximal Area of Class II Restorations
Acronym: OPUSFCLASSII
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISNFUFFBULKFGM1
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Dental Restoration Failure of Marginal Integrity
Keywords: Composite restorations; Bulk fill composites; Tooth sensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incremental Composite in Proximal Wall (Active Comparator): 38 teeth will receive class II restorations using flowable bulk fill composite to fill the cavities, leaving the proximal wall and the occlusal surface to be restored with traditional incremental composite.
  Interventions: Procedure: Restoration with Incremental Composite in Proximal Wall
- Bulk Fill Composite in Proximal Wall (Experimental): 38 teeth will receive class II restorations using flowable bulk fill composite to fill the cavities, leaving the occlusal surface to be restored with traditional incremental composite.
  Interventions: Procedure: Restoration with Bulk Fill Composite in Proximal Wall

INTERVENTIONS:
Procedure: Restoration with Incremental Composite in Proximal Wall — Proximo-occlusal lesions will receive the self-etch adhesive system Ambar Universal APS with selective acid etching, according to the manufacturers instrucions. Then, proximal wall will be completely restored with Vittra APS composite resin, using the triangular incremental traditional technique described for classe II restorations. Then, Opus Bulk Fill Flow APS will be used in the bulk technique with up to 5mm depth increments, leaving 1 mm in the occlusal for incremental Vittra APS composite resin, that will be used with the traditional incremental technique. Both composites will be light-cured with VALO light-cure unit (Ultradent, USA) for 40 seconds.
  Arms: Incremental Composite in Proximal Wall
Procedure: Restoration with Bulk Fill Composite in Proximal Wall — Proximo-occlusal lesions will receive the self-etch adhesive system Ambar Universal APS with selective acid etching, according to the manufacturers instrucions. Then, Opus Bulk Fill Flow APS resin will be used in the bulk technique with up to 5mm depth increments, leaving 1 mm in the occlusal for incremental Vittra APS composite resin, that will be used with the traditional incremental technique. Both composites will be light-cured with VALO light-cure unit (Ultradent, USA) for 40 seconds.
  Arms: Bulk Fill Composite in Proximal Wall

SUMMARY:
Treatment clinical trial, randomized, controlled, parallel, double-blinded, with two groups, that aims to evaluate the best application strategy when using a flowable bulk fill composite (Opus Bulk Fill Flow APS, FGM, Brazil) in class II cavities. Volunteers will be selected and recruited, following inclusion criteria and pre-established exclusion criteria. All volunteers will be informed and sign a term of clarification and consent. 38 enrolled patients will receive 76 Class II dental restorations, made in two different ways, one from each experimental group. Authors will perform restorations with an incremental composite (Vittra APS - FGM) associated with a bulk-fill flowable composite (Opus Bulk Fill Flow APS - FGM), in class II cavities, exposing (Group BP) or not (Group IP) the bulk fill flowable composite to the cavosurface angle on the proximal wall of the restorations. In both groups, Opus Bulk Fill Flow APS resin will be used in the bulk technique with up to 5mm depth increments, leaving 1 mm in the occlusal for incremental Vittra APS composite resin. Immediate post-operative tooth sensitivity will be evaluated after one week. Restorations will be evaluated every 6 months for pain assessment, shape, fractures, staining or recurrent caries, using FDI scores. To determine in which group each tooth will be enrolled, the authors will randomize the teeth.

DETAILED DESCRIPTION:
This is a Treatment clinical trial, randomized, controlled, parallel, double-blinded, with two groups, that aims to evaluate the best application strategy when using a flowable bulk fill composite (Opus Bulk Fill Flow APS, FGM, Brazil) in class II cavities. Volunteers will be selected and recruited, following inclusion criteria and pre-established exclusion criteria. All volunteers will be informed and sign a term of clarification and consent. All 38 enrolled patients will receive 76 Class II dental restorations, made in two different ways, one from each experimental group. All patients must have at only 20 teeth in function, must have at only 2 carious lesion in proximo-occlusal face in posterior teeth or old restorations in the same faces, with problems, that need to be changed. Those lesions must be more than 3 mm deep in occlusal area and more than 5 mm deep in at only one proximal area, should have exposed dentin, and must have at only 50% of margins in enamel. Teeth should not present periodontal mobility. Firstly, the patient will be anesthetized locally with 3% Mepivacaine solution, followed by prophylaxis with pumice powder and water. All cavities will be washed and dried after these procedures for optimal selection of color, using a color scale. Then, the rubber dam isolation of the teeth to be restored will be held. Proximo-occlusal lesions will receive the self-etch adhesive system Ambar Universal APS with selective acid etching, according to the manufacturers instrucions. Then, 2 different restorative protocols will be performed divided in two groups. Group Bulk Flow Proximal (BP): Opus Bulk Fill Flow APS resin will be used in the bulk technique with up to 5mm depth increments, leaving 1 mm in the occlusal for incremental Vittra APS composite resin, that will be used with the traditional incremental technique. Both composites will be light-cured with VALO light-cure unit (Ultradent, USA) for 40 seconds; Group Incremental Proximal (IP): Initially, proximal wall will be completely restored with Vittra APS composite resin, using the triangular incremental traditional technique described for classe II restorations. Then, Opus Bulk Fill Flow APS will be used in the bulk technique with up to 5mm depth increments, leaving 1 mm in the occlusal for incremental Vittra APS composite resin, that will be used with the traditional incremental technique. Both composites will be light-cured with VALO light-cure unit (Ultradent, USA) for 40 seconds. Immediate post-operative tooth sensitivity will be evaluated after one week. Restorations will be evaluated every 6 months for pain assessment, shape, fractures, staining, or recurrent caries, using scores. To determine in which group each tooth will be enrolled, the authors will randomize the teeth.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must have at only 20 teeth in function
* Volunteers must have at only 2 carious proximo-occlusal lesions, or old restorations that need to be changed, in different teeth
* These lesions must be more than 3 mm deep in the oclusal area and more than 5 mm deep in the proximal area, should have exposed dentin, and must have at only 50% of margins in enamel
* Teeth should not present periodontal mobility

Exclusion Criteria:

* Volunteers with periodontal disease
* Volunteers with gingival bleeding
* Volunteers that have uses anti-inflammatory drugs in the last 30 days
* Pregnant volunteers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Restoration Loss | Five years
  It will be evaluated the increase in the number of losses of dental restorations in the period of five years, verified by periodic visual clinical examination (6/6 months) based on the statement of difference of at least 25% in the amount of remaining restorations in the different groups.

SECONDARY OUTCOMES:
Marginal Pigmentation | Five years
  It will be evaluated the increase in the number of dental restorations with marginal pigmentation in the period of five years, verified by periodic clinical visual examination (6/6 months) based on the statement of difference of at least 25% in the amount of stained restorations in the different groups.
Post-Operative Hypersensitivity | Five years
  It will be evaluated the increase in the number of dental restorations with dentin hypersensitivity in the period of five years, verified by periodic clinical examination (6/6 months) based on the statement of difference of at least 25% in the amount of restorations with dentin hypersensitivity in the different groups.
Secondary Caries | Five years
  It will be evaluated the increase in the number of dental restorations with secondary caries in the period of five years, verified by periodic radiographic examination (6/6 months) based on the statement of difference of at least 25% in the amount of restorations with secondary caries in the different groups.
Marginal Adaptation | Five years
  It will be evaluated the increase in the number of dental restorations with problems in the marginal adaptation in the period of five years, verified by periodic clinical visual examination (6/6 months) based on the statement of difference of at least 25% in the amount of stained restorations in the different groups.
Color Match | Five years
  It will be evaluated the increase in the number of dental restorations with changes in the color of the restoration after clinical use, in the period of five years, verified by periodic clinical visual examination (6/6 months) based on the statement of difference of at least 25% in the amount of stained restorations in the different groups.
Proximal Contact Quality | Five years
  It will be evaluated the increase in the number of dental restorations with problems in proximal contact of the restoration after clinical use, in the period of five years, verified by periodic clinical visual examination (6/6 months) based on the statement of difference of at least 25% in the amount of stained restorations in the different groups.

CONTACTS AND LOCATIONS:
Overall Officials: MARCOS O BARCELEIRO, PhD, Study Director — Universidade Federal Fluminense
Locations (1):
- Universidade Federal Fluminense - School of Dentistry, Nova Friburgo, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chesterman J, Jowett A, Gallacher A, Nixon P. Bulk-fill resin-based composite restorative materials: a review. Br Dent J. 2017 Mar 10;222(5):337-344. doi: 10.1038/sj.bdj.2017.214. PMID 28281590
- [Background] Tardem C, Albuquerque EG, Lopes LS, Marins SS, Calazans FS, Poubel LA, Barcelos R, Barceleiro MO. Clinical time and postoperative sensitivity after use of bulk-fill (syringe and capsule) vs. incremental filling composites: a randomized clinical trial. Braz Oral Res. 2019 Sep 16;33(0):e089. doi: 10.1590/1807-3107bor-2019.vol33.0089. PMID 31531552
- [Background] van Dijken JWV, Pallesen U. Bulk-filled posterior resin restorations based on stress-decreasing resin technology: a randomized, controlled 6-year evaluation. Eur J Oral Sci. 2017 Aug;125(4):303-309. doi: 10.1111/eos.12351. Epub 2017 May 19. PMID 28524243
- [Background] van Dijken JW, Pallesen U. A randomized controlled three year evaluation of "bulk-filled" posterior resin restorations based on stress decreasing resin technology. Dent Mater. 2014 Sep;30(9):e245-51. doi: 10.1016/j.dental.2014.05.028. Epub 2014 Jun 21. PMID 24958689
- [Background] Reis A, Dourado Loguercio A, Schroeder M, Luque-Martinez I, Masterson D, Cople Maia L. Does the adhesive strategy influence the post-operative sensitivity in adult patients with posterior resin composite restorations?: A systematic review and meta-analysis. Dent Mater. 2015 Sep;31(9):1052-67. doi: 10.1016/j.dental.2015.06.001. Epub 2015 Jun 27. PMID 26122377
- [Background] Hirani RT, Batra R, Kapoor S. Comparative Evaluation of Postoperative Sensitivity in Bulk Fill Restoratives: A Randomized Controlled Trial. J Int Soc Prev Community Dent. 2018 Nov-Dec;8(6):534-539. doi: 10.4103/jispcd.JISPCD_218_18. Epub 2018 Nov 29. PMID 30596045
- [Background] da Veiga AM, Cunha AC, Ferreira DM, da Silva Fidalgo TK, Chianca TK, Reis KR, Maia LC. Longevity of direct and indirect resin composite restorations in permanent posterior teeth: A systematic review and meta-analysis. J Dent. 2016 Nov;54:1-12. doi: 10.1016/j.jdent.2016.08.003. Epub 2016 Aug 11. PMID 27523636
- [Background] Vianna-de-Pinho MG, Rego GF, Vidal ML, Alonso RCB, Schneider LFJ, Cavalcante LM. Clinical Time Required and Internal Adaptation in Cavities restored with Bulk-fill Composites. J Contemp Dent Pract. 2017 Dec 1;18(12):1107-1111. doi: 10.5005/jp-journals-10024-2184. PMID 29208783
- [Background] Guney T, Yazici AR. 24-Month Clinical Evaluation of Different Bulk-Fill Restorative Resins in Class II Restorations. Oper Dent. 2020 Mar/Apr;45(2):123-133. doi: 10.2341/18-144-C. Epub 2019 Nov 6. PMID 31693438
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. Int J Surg. 2011;9(8):672-7. doi: 10.1016/j.ijsu.2011.09.004. Epub 2011 Oct 13. No abstract available. PMID 22019563
- [Background] Costa T, Rezende M, Sakamoto A, Bittencourt B, Dalzochio P, Loguercio AD, Reis A. Influence of Adhesive Type and Placement Technique on Postoperative Sensitivity in Posterior Composite Restorations. Oper Dent. 2017 Mar/Apr;42(2):143-154. doi: 10.2341/16-010-C. Epub 2016 Nov 28. PMID 27892839
- [Background] Loguercio AD, Rezende M, Gutierrez MF, Costa TF, Armas-Vega A, Reis A. Randomized 36-month follow-up of posterior bulk-filled resin composite restorations. J Dent. 2019 Jun;85:93-102. doi: 10.1016/j.jdent.2019.05.018. Epub 2019 May 14. PMID 31100332